CLINICAL TRIAL: NCT06685796
Title: A Phase II Study of BEBT-209 in Combination With Carboplatin and Gemcitabine for the Treatment of Advanced Triple-Negative Breast Cancer
Brief Title: A Study of BEBT-209 in Combination With Chemotherapy for the Treatment of Advanced Triple-Negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BeBetter Med Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBMT-209B-P01
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Advanced Triple-Negative Breast Cancer
Keywords: BEBT-209; Safety; Efficacy; In Combination With Chemotherapy
MeSH Terms: interventions — Carboplatin; Gemcitabine; Injections

STUDY DESIGN:
Intervention Model Description: This study is designed with a total of 3 cohorts, enrolling patients with advanced triple-negative breast cancer. Subjets are randomly assigned to each cohort in a 1:1:1 ratio. Each cohort initially enrolls no fewer than 8 subjects for safety assessment, with the assessment period being the first cycle of medication (21 days). If the overall safety assessment is tolerable, the enrollment will be expanded to 30-40 subjects. During the trial, if the subjets in any of the above cohorts are unable to tolerate the treatment or there is no clinical benefit, the enrollment for that cohort will be terminated promptly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1：Carboplatin and Gemcitabine (Experimental): Carboplatin injection, dosage:AUC 2 ×(creatinine clearance rate + 25), frequency and duration of administration: administered on days 1 and 8 of each cycle, with a 21-day cycle.
  Gemcitabine hydrochloride for injection, dosage:1000mg/m², frequency and duration of administration: administered on days 1 and 8 of each cycle, with a 21-day cycle.
  Interventions: Drug: Carboplatin injection; Drug: Gemcitabine hydrochloride for injection
- Cohort 2：BEBT-209 Capsules plus Chemotherapy (Carboplatin and Gemcitabine) (Experimental): BEBT-209 Capsules, dosage: 150mg, frequency and duration of administration: administered on days 1, 2, 8, and 9 of each cycle, with a 21-day cycle. On days 1 and 8, take orally once before dinner, and on days 2 and 9, take orally once before breakfast.
  Carboplatin injection, dosage: AUC 2 × ( creatinine clearance rate + 25), frequency and duration of administration: administered on days 2 and 9 of each cycle, with a 21-day cycle.
  Gemcitabine hydrochloride for injection, dosage: 1000mg/m², frequency and duration of administration: administered on days 2 and 9 of each cycle, with a 21-day cycle.
  Interventions: Drug: BEBT-209 capsules; Drug: Carboplatin injection; Drug: Gemcitabine hydrochloride for injection
- Cohort 3：BEBT-209 Capsules plus Chemotherapy (Carboplatin and Gemcitabine) (Experimental): BEBT-209 Capsules, dosage: 150mg, frequency and duration of administration: administered on days 1, 2, 8, and 9 of each cycle, with a 21-day cycle. On days 1 and 8, take orally twice (before breakfast and before dinner), and on days 2 and 9, take orally once before breakfast.
  Carboplatin injection, dosage: AUC 2 × (creatinine clearance rate + 25), frequency and duration of administration: administered on days 2 and 9 of each cycle, with a 21-day cycle.
  Gemcitabine hydrochloride for injection, dosage: 1000mg/m², frequency and duration of administration: administered on days 2 and 9 of each cycle, with a 21-day cycle.
  Interventions: Drug: BEBT-209 capsules; Drug: Carboplatin injection; Drug: Gemcitabine hydrochloride for injection

INTERVENTIONS:
Drug: BEBT-209 capsules — BEBT-209 Capsules, dosage: 150mg, frequency and duration of administration: administered on days 1, 2, 8, and 9 of each cycle, with a 21-day cycle. On days 1 and 8, take orally once before dinner or twice (before breakfast and before dinner), and on days 2 and 9, take orally once before breakfast.
  Other Names: KCBT-0191
  Arms: Cohort 2：BEBT-209 Capsules plus Chemotherapy (Carboplatin and Gemcitabine); Cohort 3：BEBT-209 Capsules plus Chemotherapy (Carboplatin and Gemcitabine)
Drug: Carboplatin injection — Carboplatin injection, dosage: AUC 2 × (creatinine clearance rate + 25), frequency and duration of administration: administered on days 1 and 8 or days 2 and 9 of each cycle, with a 21-day cycle.
  Other Names: NSC 241240
Drug: Gemcitabine hydrochloride for injection — Gemcitabine hydrochloride for injection, dosage: 1000mg/m², frequency and duration of administration: administered on days 1 and 8 or days 2 and 9 of each cycle, with a 21-day cycle.
  Other Names: NSC 613327

SUMMARY:
This is a multicenter, open-label, two-stage Phase II clinical study to evaluate the safety and efficacy of BEBT-209 capsule in combination with carboplatin and gemcitabine for the treatment of advanced triple-negative breast cancer (TNBC).

DETAILED DESCRIPTION:
This study is designed with a total of 3 cohorts, enrolling patients with advanced triple-negative breast cancer. Subjects are randomly assigned to each cohort in a 1:1:1 ratio. Each cohort initially enrolls no fewer than 8 subjects for safety assessment, with the assessment period being the first cycle of medication (21 days). If the overall safety assessment is tolerable, the enrollment will be expanded to 30-40 subjects. During the trial, if the subjects in any of the above cohorts are unable to tolerate the treatment or there is no clinical benefit, the enrollment for that cohort will be terminated promptly.

Dosing Regimen Exploration Stage: A total of 3 cohorts are designed, namely Cohort 1, Cohort 2, and Cohort 3. Cohort 1 receives carboplatin and gemcitabine treatment, with medication administered on days 1 and 8 of each cycle, with a 21-day cycle; Cohort 2 receives BEBT-209 capsules + chemotherapy (carboplatin and gemcitabine), with medication administered on days 1, 2, 8, and 9 of each cycle, with a 21-day cycle, where on days 1 and 8, BEBT-209 capsules 150mg are administered orally only before dinner, and on days 2 and 9, BEBT-209 capsules 150mg are administered orally before breakfast on the day of chemotherapy, along with carboplatin and gemcitabine treatment; Cohort 3 receives BEBT-209 capsules + chemotherapy (carboplatin and gemcitabine), with medication administered on days 1, 2, 8, and 9 of each cycle, with a 21-day cycle, where on days 1 and 8, BEBT-209 capsules are administered orally only (150mg，twice a day, before breakfast and before dinner), and on days 2 and 9, BEBT-209 capsules 150mg are administered orally before breakfast on the day of chemotherapy, along with carboplatin and gemcitabine treatment. If the safety assessment deems the BEBT-209 dosing regimen in Cohort 2 and Cohort 3 to be intolerable, the investigators may adjust the dosing regimen design for BEBT-209 capsules.

Expansion Stage: Investigators determine the expansion cohort for a specific dosing regimen based on the combined results of safety and pharmacodynamics observed in the dosing regimen exploration stage, further exploring the safety and efficacy of BEBT-209 capsules in combination with carboplatin and gemcitabine for the treatment of advanced triple-negative breast cancer.

The study process for each subject includes three periods: the screening period, the treatment period, and the post-treatment follow-up period. The screening period lasts up to 28 days. Subjects who meet the inclusion criteria and do not meet the exclusion criteria will be enrolled to receive treatment in a 21-day treatment cycle. Hematological assessments are conducted before and after each cycle of chemotherapy, and an overall safety assessment is conducted according to the protocol during the study period; after the first dose during the treatment period, the first two tumor assessments are conducted every 9 weeks, and from the third assessment onward, every 12 weeks. Participants can continue to receive the study medication until disease progression (PD), death, intolerable toxicity, or withdrawal of informed consent (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years old, female;
2. The subject has fully understood and is willing to sign the Informed Consent Form (ICF);
3. Confirmed diagnosis of HR-negative, HER2-negative locally recurrent or metastatic breast cancer by pathological biopsy;
4. Estrogen and progesterone receptor immunohistochemical assessment of tumor tissue is negative (defined as <1% nuclear staining), and HER2 is negative (i.e., no overexpression, including local immunohistochemical assessment [0 or 1+], or immunohistochemical assessment [2+] with negative in situ hybridization testing);
5. The subject has previously received 1-2 lines of systemic treatment (if progression within 12 months after the last treatment of adjuvant/new adjuvant, it can be considered as one line of treatment);
6. At least one measurable lesion in accordance with Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria;
7. Eastern Cooperative Oncology Group (ECOG) score of 0-1 , and no decline in physical performance in the past two weeks;
8. Life expectancy of at least 12 weeks;
9. Adequate organ and bone marrow function, defined as follows:

   1. Absolute neutrophil count (ANC) ≥ 1500/mm³ (1.5 × 10^9/L);
   2. Platelets ≥ 100,000/mm³ (100 × 10^9/L);
   3. Hemoglobin ≥ 9 g/dL (90 g/L);
   4. Alanine Aminotransferase (ALT) or Aspartate Transaminase (AST) both ≤ 2.5 × ULN, when liver metastasis is present, ALT or AST both ≤ 5.0 × Upper limit of normal value (ULN);
   5. Total bilirubin (TBIL) ≤ 1.5 × ULN, when liver metastasis is present, ≤ 3.0 × ULN;
   6. Serum creatinine ≤ 1.5 × ULN or estimated creatinine clearance ≥ 60 mL/min (based on the Cockcroft and Gault formula);
10. All acute toxic reactions from previous anticancer treatments or surgical procedures have resolved to baseline severity or National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 ≤ Grade 1 (except for alopecia or other toxicities that the investigator deems have no safety risk to the patient);
11. Women of childbearing age must have a negative serum pregnancy test within 7 days prior to the start of study medication, and must be willing to use a medically recognized, highly effective contraceptive method (such as intrauterine device, birth control pills, or condoms) during the study period and for one month after the last administration of the study medication.

Exclusion Criteria:

1. Previous treatment with gemcitabine;
2. Previous treatment with carboplatin for locally recurrent unresectable or metastatic breast cancer is allowed if it was administered in the adjuvant or neoadjuvant setting more than 6 months before the first metastatic relapse;
3. Concurrent central nervous system metastases or leptomeningeal disease requiring immediate radiotherapy or corticosteroid treatment; patients must discontinue steroid medication for at least 14 days before the first administration of the study drug. No stereotactic radiosurgery within 7 days or whole brain radiotherapy within 14 days before the first administration of the study drug;
4. Previous receipt of hematopoietic stem cell or bone marrow transplantation;
5. Within 7 days prior to study entry, the patient has received the following treatments:

   1. Medications known to be strong inhibitors/inducers of CYP3A4;
   2. Medications known to significantly prolong the QT interval or cause torsades de pointes (antiarrhythmic drugs such as quinidine, disopyramide, procainamide, sotalol, etc.);
6. Within 14 days prior to study entry, the patient has received radiotherapy, or within 21 days prior to study entry, the patient has received other investigational drug treatment or cytotoxic chemotherapy;
7. Known history of hypersensitivity or suspected allergic symptoms to any component of BEBT-209, carboplatin, or gemcitabine;
8. In a resting state, the average corrected QT interval (QTc) obtained from 3 Electrocardiogram (ECG) examinations is >480msec (corrected using the Fridericia method); history of long QT syndrome or confirmed family history of long QT syndrome; history of clinically significant ventricular arrhythmias, or current use of antiarrhythmic drugs or implantation of defibrillation devices for the treatment of ventricular arrhythmias;
9. Uncontrolled electrolyte disturbances that may affect the action of QTc-prolonging drugs (such as hypocalcemia <1.0mmol/L, hypokalemia < lower limit of normal, hypomagnesemia <0.5mmol/L), but re-screening is allowed after interventional treatment;
10. History of myocardial infarction, severe/unstable angina, persistent arrhythmias ≥ Grade 2 according to NCI CTCAE version 5.0, any grade of atrial fibrillation, coronary/ peripheral artery bypass surgery, symptomatic congestive heart failure, cerebrovascular accident (including transient ischemic attack or symptomatic pulmonary embolism);
11. Active inflammatory bowel disease or chronic diarrhea, short bowel syndrome, or any upper gastrointestinal surgery including gastrectomy; known malabsorption syndrome or other conditions that may impair the absorption of BEBT-209;
12. Clinically significant active infections, including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related diseases. Active hepatitis B is defined as positive for hepatitis B surface antigen (HBsAg) or hepatitis B e antigen (HBeAg), and HBV-DNA greater than the upper limit of normal for the research center. Patients with quantitative HBV DNA greater than the upper limit of normal for the research center are allowed to receive antiviral treatment before screening to reduce the viral load to within the normal range, but must continue to receive antiviral treatment for hepatitis B during the trial; active hepatitis C is defined as HCV RNA above the detection limit;
13. Diabetes with poor blood sugar control as judged by the investigator;
14. Women who plan to conceive again within 5 years without having undergone oocyte cryopreservation;
15. Recent or active suicidal ideation or behavior;
16. Currently participating in or about to participate in other interventional clinical trials;
17. Other serious acute or chronic medical or psychiatric conditions or laboratory test abnormalities that may increase the risk of participating in the study or the risk associated with the administration of the study drug, or interfere with the study results, and any other conditions that the investigator deems the patient is not suitable to participate in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Progression-free survival
AE | From the first administration of the study drug to 28 days after the last administration of the study drug
  Adverse event

SECONDARY OUTCOMES:
OS | From date of administration until date of death from any cause,assessed up to 24 months.
  Overall survival
ORR | During the treatment period, the first two assessments are conducted every 9 weeks, and starting from the third assessment, they are conducted every 12 weeks,assessed up to 24 months.
  Objective response rate
DCR | During the treatment period, the first two assessments are conducted every 9 weeks, and starting from the third assessment, they are conducted every 12 weeks,assessed up to 24 months.
  Disease control rate
TTR | During the treatment period, the first two assessments are conducted every 9 weeks, and starting from the third assessment, they are conducted every 12 weeks,assessed up to 24 months.
  Time to response
DOR | During the treatment period, the first two assessments are conducted every 9 weeks, and starting from the third assessment, they are conducted every 12 weeks,assessed up to 24 months.
  Duration of Response

CONTACTS AND LOCATIONS:
Overall Officials: Quchang Ouyang, Phd, Principal Investigator — Hunan Cancer Hospital; Qiang Liu, Phd, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (2):
- China (2):
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Hunan Cancer Hospital, Changsha, Hunan